CLINICAL TRIAL: NCT05365594
Title: Biomechanical Analysis of Gait in a Walking Boot With Contralateral Foot Lift
Brief Title: Biomechanical Analysis of CAM Boot and EVENUp Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202102519
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Biomechanics; Limb Length Discrepancy
Keywords: CAM Boot; EVENup

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Self Selected Pace (Active Comparator): Tennis shoes, CAM Boot, CAM Boot plus EvenUp Lift
  Interventions: Device: Controlled Ankle Movement Boot; Device: EVENUp Lift
- Speed Walking Pace (Active Comparator): Tennis shoes, CAM Boot, CAM Boot plus EvenUp Lift
  Interventions: Device: Controlled Ankle Movement Boot; Device: EVENUp Lift

INTERVENTIONS:
Device: Controlled Ankle Movement Boot — Walking boot used for orthopaedic foot injuries
Device: EVENUp Lift — Orthotic shoe lift worn on contralateral foot to increase leg length
  Other Names: Foot Lift

SUMMARY:
Walking boots are a common form of durable medical equipment Orthopaedic surgeons prescribe both post-operatively and in the treatment of lower extremity injuries. Walking boots create a limb length discrepancy (LLD) which effects joint angles and moment arms in the lower extremities and the spine. These altered mechanics lead to reported back, hip, and knee pain in patients who are prescribed walking boots. Current walking boot literature evaluates gait and ground reaction forces (GRF), focusing primarily on the lower extremities, neglecting the remainder of the kinetic chain including the spine. Alternatively, there is a body of literature evaluating the effects of congenital LLD on spine and posture. However, there is paucity in the literature reporting both the effects of a walking boot on the entire kinematic chain and the subsequent effects of a corrective foot lift. The investigators seek to evaluate lower extremity and spinal kinematics using a motion analysis capture system with healthy subjects undergoing walking trials while wearing normal shoes, a walking boot, and a walking boot with contralateral foot lift. The investigators hypothesize a corrective foot lift will decrease the asymmetrical effects of a walking boot, recreating the kinematics of a more normal gait.

DETAILED DESCRIPTION:
The goal of this study is to understand the kinematic effects of a walking boot on joint angles, moment arms and ground reaction forces in the spine and lower extremities. Additionally, the investigators will examine the effects a corrective foot lift, EVENup, has on these variables. This goal will be accomplished through (2) aims:

Aim 1. Compare the differences in kinetics and kinematics of the spine and lower extremities during normal gait and wearing a walking boot.

Aim 2. Compare spine and lower extremity kinetics and kinematics differences in a walking boot with and without the use of a corrective foot lift on contralateral leg.

Hypothesis: A contralateral foot lift will significantly reduce the altered mechanics created by a walking boot. These results would encourage physicians to recommend a contralateral foot lift when prescribing a walking boot to decrease secondary site pain.

Methodology: All subjects will participate in a gait analysis session in which their joint kinematics and kinetics will be recorded using skin-marker motion capture and treadmill force plates. Skin-marker motion capture involves placing reflective markers on palpable bony landmarks, such as the medial and lateral malleoli. These reflective markers are secured to the subject's skin using adhesive tape. Specialized, infrared cameras are then used to record the location of these markers as the subject walks at a self-selected speed and a specified speed denoted as faster pace. A self-selected speed will be determined by slowing increasing the speed of the treadmill until the subject feels like they are walking at a comfortable everyday speed. The faster pace will be determined by having the subject walk as if they are speed walking.

Participants will complete two trials with 3 different scenarios in each trial : 1) treadmill walking with regular shoes, 2) treadmill with walking boot and 3) treadmill with walking boot and corrective lift. Each participant's trial order will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cohort:
* Age of 18 to 40 years
* No history of lower extremity injury in last 5 years
* No history of lower limb discrepancy

Exclusion Criteria:

* Pregnant women; minors (under age 18); mentally disabled; any persons incarcerated, on parole, on probation, or awaiting trial.
* Persons with medical history of spinal, hip, or other musculoskeletal pathology that may alter walking mechanics.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Compare the differences in kinetics and kinematics of the spine during normal gait and wearing a walking boot | Day 1
  Take range of motion measurements of the spine

SECONDARY OUTCOMES:
Compare spine kinetics and kinematics differences in a walking boot with and without the use of a corrective foot lift on contralateral leg | Day 1
  Take range of motion measurements of the spine
Compare the differences in kinetics and kinematics of the lower extremities during normal gait and wearing a walking boot | Day 1
  Take range of motion measurements of the knee
Compare the differences in kinetics and kinematics differences in a walking boot with and without the use of a corrective foot lift on contralateral leg | Day 1
  Take range of motion measurements of the knee

CONTACTS AND LOCATIONS:
Overall Officials: Michael Talerico, MD, Principal Investigator — University of Florida
Locations (1):
- UF & Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No